CLINICAL TRIAL: NCT05950958
Title: The Impact of Audio and Visual Intervention in Preventing ICU Delirium in Critically Ill Patients : A Randomized Clinical Trial
Brief Title: Prevention of Delirium in ICU Using Multimodal Interventions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ho Geol Ryu, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Delirium_ICU
Record Dates: First submitted 2022-07-28; First posted 2023-07-18 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Intensive Care Unit Delirium
Keywords: Delirium; Intensive Care Unit; Non-pharmacological intervention
MeSH Terms: conditions — Delirium | interventions — Combined Modality Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal therapy group (Experimental): Continuous regional cerebral oxygen saturation and processed electroencephalogram (EEG) are monitored.
  Multimodal therapy with conventional care are provided to prevent delirium. Ongoing orientation: 3 times per day Sensory correction: the hearing device and the glasses are supplied. Cognitive stimulation: a portable monitor is used to provide visual stimulation, and a directional speaker is used to avoid disturbing the alarm of the patient's life supportimng system.
  Sleep promotion: the lights are turned off from 10 pm to 7 am, and the indirect light source is used if necessary.
  Interventions: Other: Multimodal therapy for prevention of delirium
- Conventional care group (No Intervention): Continuous regional cerebral oxygen saturation and processed electroencephalogram (EEG) are monitored.
  Conventional care: If sedation is required, dexmedetomidine is considered as the first-line sedative drug. The sedation is interrupted daily and the possibility of awakening is assessed. Pain with NRS score above 3, is controlled with opioid.
  For patients with Richmond Agitation Sedation Scale (RASS) -4 or -5, possible items are provided.

INTERVENTIONS:
Other: Multimodal therapy for prevention of delirium — Multimodal therapy for prevention of delirium
  Arms: Multimodal therapy group

SUMMARY:
This study was designed to evaluate the impact of non-pharmacological multimodal interventions including ongoing orientation, sensory correction, setting of familiar circumstance and promotion of sleep enviromnet for prevention of delirium in intensive care unit.

DETAILED DESCRIPTION:
Delirium significantly increases not only the length of the intensive care unit stay and overall mortality, but also the likelihood of persistant cognitive impairment after recovery. However there is no definitive treatment for delirium, thereby it is important to prevent delirium before it occur. Researches also have focused on the prevention of delirium or the reduction of duration of delirium.

Several studies evaluated the effect of non-pharmacological treatment, such as improvement of orientation, prevention of sensory deprivation, active pain control and prevention of dehydration, to reduce the occurrence of delirium and the results were inconsistent depending on the patients included. However, there have been no randomized clinical trials that have tested the effect of prevention of delirium by applying non-pharmacological multimodal approaches in the intensive care unit for Korean patients.

A randomized controlled trial was planned to evaluate the impact of on-pharmacological multimodal interventions including ongoing orientation, sensory correction, setting of familiar circumstance and promotion of sleep enviromnet for prevention of delirium in intensive care unit in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 50 years who are expected to spend more than 24 hours in the intensive care unit

Exclusion Criteria:

* Patients who developed delirium before entering the intensive care unit
* Patients with cognitive impairment
* Patients who have hearing or vision deficits, or have difficulty in communication
* Patients who are expected to die within 24 hours or do not want life-sustaining treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with delirium | From ICU admission up to day 28 or discharge from ICU or death
  Delirium assessed by Confusion Assessment Method for the ICU (CAM-ICU)

SECONDARY OUTCOMES:
Delirium-free days | From ICU admission up to day 28 or discharge from ICU or death
  Delirium assessed by Confusion Assessment Method for the ICU (CAM-ICU)
Severity of delirium | From ICU admission up to day 28 or discharge from ICU or death
  Confusion Assessment Method for the ICU-7 (CAM-ICU-7) delirium severity score
Accidental extubation or disconnection of treatment devices | From ICU admission up to day 28 or discharge from ICU or death
  Accidental extubation or disconnection of treatment devices
ICU and hospital length of stay | From ICU admission up to day 28 or discharge from ICU or death
  Duration of ICU and hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Ho Geol Ryu, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No